CLINICAL TRIAL: NCT04582773
Title: Improving the Outcomes of Community-based Management of Acute Malnutrition
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Alliance for International Medical Action (Other); University of Maiduguri Teaching Hospital (Unknown); Tampere University (Other)
Responsible Party: Principal Investigator, Christopher Parshuram, Principal Investigator, The Hospital for Sick Children
Other Study IDs: REB1000063224
Record Dates: First submitted 2020-09-08; First posted 2020-10-12 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe acute malnutrition (SAM) affects 16 million children at any one time and is responsible for the deaths of over 500,000 children under 5 years of age each year. Treatment for severe acute malnutrition is based on the Community-based Management of Acute Malnutrition (CMAM) model. The current methods used for detecting high risk children have not prevented 5% mortality observed in regions using this program. The purpose of the study is to provide evidence that objective methods for detecting high risk children can be used to optimize efficiency of Community-based Management of Acute Malnutrition (CMAM) treatment programs and thus improve child health outcomes.

DETAILED DESCRIPTION:
A prospective observational study in inpatient care within community-based management of acute malnutrition(CMAM) program run by the nongovernmental organization called Alliance for International Medical Action (ALIMA) within the University of Maiduguri Teaching Hospital, Maiduguri, Nigeria

The objectives of the study are to validate the BedsidePEWS scores as a measure of severity of illness in children who are treated as inpatients for severe acute malnutrition and to compare the BedsidePEWS scores with other risk factors associated for mortality and relapse of children with severe acute malnutrition. The design is a prospective observational study of 1000 children admitted as inpatients in a CMAM program in Maidaguri Teaching Hospital in Maidaguri, Nigeria. Data collection (estimated duration 4-5 months) involves vital signs, and risk factor assessment every 12 hours for duration of hospitalization. Blood test for hemoglobin and malaria will be done once upon admission. Outcomes will be measured every 12 hours and include mortality and/or escalation and de-escalation of care. Logistic regression with significance testing will be used to compare BedsidePEWS scores and risk factors between patients and among individual patients within the outcome categories. Exploratory sensitivity analyses will repeat the main logistic regression analyses to evaluate the performance of partial BedsidePEWS score in patients with missing data of 1-3 of the 7 components, by randomly removing 1-3 data elements from the score calculation from patients, and by removing systolic blood pressure from scoring.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 to 59 months
* Diagnosed with severe acute malnutrition (criteria for severe acute malnutrition is <3Z Weight for Height Z score, and/or MUAC <115mm, and/or bilateral pitting oedema)
* Meet the criteria for admission into inpatient care (failed appetite test, and/or medical conditions).

Study amendment for inclusion: children with and without severe acute malnutrition admitted to emergency pediatric unit (EPU)

Exclusion Criteria:

- Children with congenital anomalies that interfere with feeding (ie. cleft lip and/or palate); previous enrolment in this study.

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 1-59 months with severe acute malnutrition admitted into inpatient care within CMAM program run by the non-governmental organization called Alliance for International Medical Action (ALIMA) within the University of Maiduguri Teaching Hospital, Maiduguri, Nigeria
Sampling Method: Non-Probability Sample
Enrollment: 1087 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Inpatient mortality | From admission to inpatient care until the the earlier of the date of discharge from inpatient care or ten weeks after enrolment
  survival or death during inpatient care

SECONDARY OUTCOMES:
Number of Children receiving inpatient care who required escalation of treatment | From admission to inpatient care until the the earlier of the date of discharge from inpatient care or ten weeks after enrolment
  transfer from unit of lower to higher level of care within inpatient treatment
Number of Children receiving inpatient care who required de-escalation of treatment | From admission to inpatient care until the the earlier of the date of discharge from inpatient care or ten weeks after enrolment
  transfer from unit of higher to lower level of care within inpatient treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chris Parshuram, MD/PHD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- University of Maiduguri Teaching Hospital, Maiduguri, Borno State, Nigeria